CLINICAL TRIAL: NCT00062907
Title: Phase I Open-Label Dose Escalation Trial Evaluating The Safety And Immunogenicity Of Sequential Administration Of Recombinant DNA And Adenovirus Expressing L523S Protein In Patients With Early Stage Non-Small Cell Lung Cancer
Brief Title: Safety and Immunogenicity of Recombinant DNA and Adenovirus Expressing L523S Protein in Early Stage Non-Small Cell Lung Cancer
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Corixa Corporation (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCL5001-01
Record Dates: First submitted 2003-06-17; First posted 2003-06-19 (Estimated); Last update posted 2006-12-06 (Estimated); Status verified 2004-11

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

INTERVENTIONS:
Biological: Recombinant DNA- pVAX/L523S
Biological: Recombinant adenovirus- Ad/L523S

SUMMARY:
The purpose of this trial is to examine the safety and immunogenicity of a therapeutic vaccine regimen with recombinant DNA and adenovirus expressing L523S protein in patients with early stage non-small cell lung cancer. The vaccine regimen will consist of two fixed doses of recombinant DNA (pVAX/L523S) followed by two doses of recombinant adenovirus (Ad/L523S). The trial will evaluate the dose escalation of Ad/L523S through three cohorts of patients.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the safety of the vaccine regimen administered as two doses of pVAX/L523S and two doses of Ad/L523S.

The secondary objectives of the study are:

* To provide initial evidence as to whether CD8+ and CD4+ T cell responses specific for L523S protein can be elicited by two doses of pVAX/L523S followed by two doses of Ad/L523S
* To provide initial evidence as to whether antibody responses specific for L523S protein can be elicited by two doses of pVAX/L523S followed by two doses of Ad/L523S
* To investigate the extent to which dose escalation of Ad/L523S affects the elicited immune response

ELIGIBILITY:
INCLUSION CRITERIA:

* Histologically and surgical confirmed diagnosis and stage of IB, IIA, or IIB non-small cell lung cancer (NSCLC) according to the Revised International System for Staging Lung Cancer
* Primary surgical resection of lung cancer greater than or equal to 4 weeks and less than or equal to 3 years prior to the Day 0 visit
* No evidence of disease by standard diagnostic tests
* Chest X-ray and physical examination showing no active disease
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1
* WBC count greater than or equal to 3,000 cells/mm3 and ANC greater than or equal to 1,500 cells/mm3
* Hemoglobin value greater than or equal to 10.0 g/dL and a platelet count greater than or equal to 125,000 cells/mm3
* Adequate renal function (defined as serum creatinine <1.5 times the upper limit of normal for females and males)
* Normal hepatic function (defined as serum bilirubin <1.5 times the upper limit of normal, AST <2.5 times the upper limit of normal and alkaline phosphatase <1.5 times the upper limit of normal)
* Ability to understand and willingness to sign an IRB-approved written consent prior to study enrollment
* Female patients must be greater than or equal to 60 years of age, or greater than or equal to 5 years amenorrhea or surgically sterile
* Male patients who are capable of fathering a child and whose partners are capable of having a child must agree to use adequate contraception for 6 months after enrollment (for men or women-surgical sterilization; for women-hormonal contraceptives, vaginal ring or IUD)
* Absolute CD4+ cell count of >200 cells/mm3

EXCLUSION CRITERIA:

* Received pre- or post-operative radiotherapy
* Received prior biologic, immunologic, or gene therapy for cancer
* Received an investigational drug (new chemical entity) within three months of study entry
* Received antibiotics within 2 weeks of Day 0 visit
* Received systemic or inhaled corticosteroids or immunosuppressive therapy within 4 weeks of Day 0 visit (Use of topical corticosteroids and/or eye drops containing glucocorticosteroids is acceptable)
* History of active autoimmune diseases such as, but not limited to, systemic lupus erythematosis, sarcoidosis, rheumatoid arthritis, glomerulonephritis, vasculitis, or inflammatory bowel disease
* History of bleeding in stools and/or diarrhea within 4 weeks of Day 0 visit
* History of anaphylaxis or severe allergic reaction to vaccines or unknown allergens
* Received any commercial vaccine within 2 weeks of Day 0 visit
* Received a major organ allograft
* Current or previous diagnosis of paraneoplastic syndrome
* Evidence of a clinically significant active pulmonary infection, emphysema, FeV1 less than or equal to 50% predicted, DLCO less than or equal to 50% predicted, pulse oximetry less than or equal to 92% at the time of study entry
* Known to be HIV positive
* Results of virology screening indicate positive serology for HCV (hepatitis C virus) and/or HBsAG (hepatitis B surface antigen). Positive serology for HBV antibodies is allowed.
* History of other malignancies at other sites, except effectively treated non-melanoma skin cancers, superficial bladder cancer or carcinoma in situ of the cervix or an effectively treated malignancy that has been in remission for greater than 5 years and is highly likely to have been cured
* Uncontrolled medical problems (neurological, cardiovascular, gastrointestinal, genitourinary or other illness) considered as unwarranted high risk for investigational new drug treatment
* Patient is lactating
* Staging classification of TX or NX or MX
* Prior adjuvant chemotherapy within 8 weeks prior to the Day 0 visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9
Dates: Start 2003-05

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Cancer Centers of Florida, Ocoee, Florida
  - Mary Crowley Medical Research Clinic, Dallas, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Swedish Cancer Institute, Seattle, Washington
  - Cancer Care Northwest, Spokane, Washington